CLINICAL TRIAL: NCT02223624
Title: Effect of an Eccentrically Biased Aerobic Exercise Program on Quality of Life and Functional Capacity in People With Chronic Heart Failure: A Randomized Controlled Trial.
Brief Title: Effect of an Eccentric Exercise Program on Quality of Life and Function in People With Chronic Heart Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: La Trobe University (Other)
Collaborators: Northern Hospital, Australia (Other)
Responsible Party: Principal Investigator, Rachel Ellis, Clinical Leader Physiotherapist, La Trobe University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: LR49.2013 FHEC13/260 LaTrobeU; LR 49.2013 (Other: Northern Health)
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Chronic Heart Failure
Keywords: eccentric; exercise; heart disease; chronic heart failure; rehabilitation
MeSH Terms: conditions — Motor Activity; Heart Diseases | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- eccentric aerobic exercise group (Experimental): Eccentric aerobic exercise group: Participants in this group will participate in an eccentric aerobic exercise rehabilitation program for a total of eight weeks, two sessions per week. Outcome measurements will be taken post exercise program and also after a 3 month follow-up period. Each session will be approximately 60 minutes in duration and include approximately 10 minutes of warm up (stretches), eccentric stepper aiming for 20 minutes, walking and light weights, followed by a five minute cool-down period.
  Interventions: Other: walking and light weights; Other: eccentric aerobic exercise
- Concentric aerobic exercise group (Active Comparator): Concentric aerobic exercise group (usual care): The length of the concentric aerobic exercise based rehabilitation program will be the same as the study group- twice weekly exercise sessions for 8 weeks. Outcome measurements will also be taken after a 3-month follow-up period.
  Participants in the concentric aerobic exercise group will participate in the same warm-up and cool down period as the eccentric group. They will also complete walking and light weights. To replace the 20 minutes of eccentric exercise, concentric participants will complete approximately 20 minutes of exercise bike, stair climbing and rowing as able with required rests.
  Interventions: Other: walking and light weights; Other: concentric aerobic exercise
- Waiting list control (No Intervention): Waiting list (no exercise): Participants assigned to this group will not receive any intervention during the study period. They will be assessed like other participants at baseline and after eight weeks, but not at three-month follow-up due to ethical concerns around withholding care known to be effective. Given that there is a waiting list for the current exercise program of 4-12 weeks, it is felt that delaying care for a set period of eight weeks is not of ethical concern. Following the completion of assessments, waiting list participants will be able to complete the traditional exercise program as usual but not as participants of the study's experimental groups.

INTERVENTIONS:
Other: walking and light weights
  Arms: Concentric aerobic exercise group; eccentric aerobic exercise group
Other: eccentric aerobic exercise
  Arms: eccentric aerobic exercise group
Other: concentric aerobic exercise
  Arms: Concentric aerobic exercise group

SUMMARY:
Many studies have shown that exercise training is beneficial for patients with chronic heart failure (CHF). Heart Foundation guidelines strongly recommend regular physical activity and referral to a specifically designed rehabilitation program for all patients with CHF who are medically stable. Such programs usually comprise aerobic exercises such as walking, and light weightlifting with care to avoid heavy straining due to stress that this may place on the heart.

Eccentric contractions are those in which the muscle lengthens as it contracts. Exercise involving eccentric contractions is known to increase muscle strength and this type of exercise also requires less oxygen. This is because it requires less power to resist lowering a weight than it does to lift a weight. Initial evidence suggests that this form of exercise has favourable outcomes in the frail elderly and those with chronic disease.

This study aims to determine if eccentric exercise can be applied to patients with heart failure to increase their physical function while using less energy so that exercise is more tolerable for patients who complain of significant breathlessness and fatigue. This study also aims to determine if eccentric exercise is a safe alternative exercise option for patients at risk of negative events.

The investigators propose to run a randomised controlled trial. Eccentric exercise will be delivered to a group of heart failure patients referred to the existing heart failure rehabilitation program at the Northern Hospital. The program will consist of eight weeks of twice weekly exercise of one hour's duration comprising eccentric exercise combined with walking and light weight training. This will be compared to a group of patients participating in the current exercise program consisting of light weightlifting and aerobic exercises for the same length and duration of exercise and also to a third group of patients who will be wait listed for 8 weeks. Following the completion of the eight week waiting period, these patients will be offered the option of joining the standard exercise program.

The investigators expect that the eccentric exercise group will have improved walking capacity and quality of life compared with the traditional program and the wait-list control group. It is also possible that there is no difference between the eccentric and traditional program in terms of functional outcomes but that the participants report that eccentric exercise is easier.

DETAILED DESCRIPTION:
BACKGROUND A systematic literature review we conducted yielded two trials investigating eccentric exercise in patients with coronary artery disease and two trials in the chronic heart failure population. Eccentric exercise was reported to be a safe form of exercise for coronary patients, causing minimal heart and breathing stress and being perceived as "fairly light" exertion. Eccentric exercise, when compared with concentric exercise (shortening contractions) resulted in comparable improvements in muscle strength and walking distance, often with reduced oxygen usage.

With no increase in negative events with coronary patients, recently eccentric exercise has been trialed in heart failure patients. One trial looked at six-minute walk test differences in patients with mild heart failure following a program of eccentric or concentric cycling. They found that although both groups improved their walking distance, the eccentric exercise was completed at lower levels of work and stable heart rates. A second trial completed eccentric exercise by descending stairs, compared with participants who climbed stairs and measured knee muscle strength. They reported that participants found the stair descending easy with significant improvements in static strength but not eccentric (lengthening) or concentric (shortening) force. Both of these studies were limited by a population of a small number (12-15) of participants primarily males, with poorly defined or mild heart failure.

RESEARCH AIMS Given the limited evidence in coronary patients and more specifically heart failure patients, this current study aims to fill knowledge gaps by looking at the effects of eccentric exercise on both males and females, with mild to moderate heart failure, of both heart failure types- systolic (heart contraction problems) and diastolic (heart relaxation problems). We aim to include measures of both function and quality of life. We will also monitor compliance and patient satisfaction with the aim of developing a safe and tolerable exercise program that is feasible for implementation in heart failure rehabilitation programs.

METHODS Participants will be recruited through The Northern Hospital heart failure outpatient medical clinics and also through referral to the current rehabilitation program following inpatient admission or G.P referral. This study will be a prospective, three-armed, parallel-design, randomised controlled trial with a 1:1:1 ratio. A separate randomisation procedure will be prepared for each of the three included New York heart association heart failure classes so that disease severity will not affect the results.

As well as the primary outcomes of walking capacity and quality of life, secondary outcomes will include lower limb strength and levels of fatigue. We will also monitor adherence, attendance, pain, and any adverse events occurring in any session.

Demographic and outcome data will be analysed for between group differences at baseline. To determine whether group 1 improved more than groups 2 and 3 immediately after the 8-week program, data will be analysed with analysis of covariance using the baseline measures as covariates. Categorical outcome variables (death or hospital admission) will be analysed with relative risk ratios. To avoid bias and to maximise the randomisation process, intention to treat analysis will be utilised. Participants withdrawing from the project will be followed up where possible. Where data are missing, the carry forward technique will be used, which assumes that missing data remain constant. Finally, correlations between the secondary outcome variables and the primary outcome variables will also be examined to detect where associations exist as well as associations between outcomes and types of heart failure (systolic or diastolic). Significance level of P<.05 will be used for hypotheses testing.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years
* a clinical diagnosis of heart failure either systolic or diastolic on transthoracic echocardiogram
* mild to moderate heart failure
* medically stable heart failure
* have received approval when assessed by the group physiotherapist to participate in the exercise program as is usual practice. Where concerns arise during assessment, clearance will be sought from the treating cardiologist.

Exclusion Criteria:

* hospitalisation for a CHF exacerbation within the previous month
* severe heart failure classified as level four on the New York heart association classification (short of breath at rest)
* unstable medical condition such as uncontrolled angina, diabetes or hypertension
* dementia or a psychological disorder that would interfere with participation in group exercise
* participation in a cardiac or heart failure rehabilitation program in the prior six months
* contraindications to exercise (ie aneurysm, valvular disease)
* the presence of any pre-existing neurological or musculoskeletal condition, for example stroke, that on assessment is deemed to interfere with exercise participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
functional improvement measured by change in six-minute walk distance | post 8-week exercise program and 3-month follow-up

SECONDARY OUTCOMES:
Quality of life measured by participant questionnaire | post 8-week exercise program and 3-month follow-up

OTHER OUTCOMES:
Fatigue as measured by participant questionnaire | post 8-week exercise program and 3-month follow-up
lower limb strength as measured as a one-repetition maximum leg press | post 8-week exercise program and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rachel E Ellis, Principal Investigator — Northern Hospital, Australia; Kwang Lim, Principal Investigator — Melbourne Health; Karen J Dodd, Principal Investigator — Victoria University; Anne E Holland, Principal Investigator — La Trobe University; Nora Shields, Principal Investigator — La Trobe University
Locations (1):
- The Northern Hospital, Epping, Victoria, Australia

REFERENCES:
- [Derived] Ellis RE, Dodd KJ, Holland AE, Lim K, Tacey M, Shields N. Effect of eccentric exercise on quality of life and function in people with chronic heart failure: a pilot randomised controlled trial. Disabil Rehabil. 2022 Jun;44(12):2705-2714. doi: 10.1080/09638288.2020.1836679. Epub 2020 Nov 11. PMID 33174464